CLINICAL TRIAL: NCT02311374
Title: Human Brain Mapping of the Apparent Diffusion Coefficient (ADC) During Sleep and Wakefulness
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 150031; 15-AA-0031
Record Dates: First submitted 2014-12-05; First posted 2014-12-08 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-07-29

CONDITIONS: Brain Mapping
Keywords: Human Brain; Sleep; EEG; Magnetic Resonance Imaging (MRI); Apparent Diffusion Coefficient (ADC)
MeSH Terms: interventions — Functional Status; Brain Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 2 (Sham Comparator): ADC will be measured in the same subject in the wake state (following a night of regular sleep) and during sleep (following a night of sleep deprivation). The MRI scans will be done in the morning (9-12 pm), once while the subject is sleeping (following a night of sleep deprivation) and once while awake (following regular sleep 9 AM-12 PM).
  Interventions: Other: Brain connectivity and physiology; Other: Brain Wave
- Phase I (Sham Comparator): ADC will be measured in the same subject in the wake state (following a night of regular sleep) and during sleep (following a night of sleep deprivation). The MRI scans will be done in the morning (9 AM-12 pm), once while the subject is sleeping (following a night of sleep deprivation) and once while awake (following regular sleep 9 AM 12 PM).
  Interventions: Other: Brain connectivity and physiology; Other: Brain Wave

INTERVENTIONS:
Other: Brain connectivity and physiology — Two MRI scanning session will be obtained for each participant both at the same time of day (9AM 12 PM). In one occasion they will be scanned after a night of rested sleep while awake and on another day they will be scanned after one night of sleep deprivation while sleeping in the scanner. In addition to the most sensitive technique selected in the development phase (either DWI or MT), each imaging MRI session will include (1) a resting-state functional connectivity (RSFC; 10 minutes) scan using single-shot T2*-weighted EPI; and (2) quantitative T1 relaxometry (T1) in a CSF voxel (1mL; cubic) using an inversion recovery experiment with increased interpulse intervals (TI = 200, 300, 400, 500, 700, 1000, 1500, 2000, 3000, 5000, 10000 ms) and a long TR (10000 ms; scan time 2 min) to assess the level of solutes in CSF.
Other: Brain Wave — ECG will be used to monitor heart rate variability (HRV), which differ significantly between the waking state and the different sleep stages

SUMMARY:
Background:

- The glymphatic system helps keep harmful waste from building up in the brain. Researchers think it is more active in people during sleep than while awake. They want to study the glymphatic system using magnetic resonance imaging (MRI).

Objective:

- To see if there are differences in the way waste is removed from the brain while a person is sleeping versus awake.

Eligibility:

- Healthy people age 18-60.

Design:

* This study is in 2 parts.
* For the technical part (discontinued), participants will be screened with medical history and physical exam. They will have urine and breath alcohol tests.
* Participants will have 2 MRI scans. Before the scans, they will have urine and breath alcohol tests, and complete a questionnaire.
* For MRI, participants will lie on a table that slides in and out of a metal cylinder. A device will be placed over their head. They will lie still for up to 20 minutes at a time. They may be asked to stay awake or fall asleep for up to 2 hours at a time.
* For the research part, participants will be screened with medical history and physical exam. They will have urine and breath alcohol tests. For 1 week they will wear a device that monitors their activity and sleep.
* Participants will stay at NIH overnight. They will give a blood sample, have urine and breath alcohol tests, and complete a questionnaire.
* Participants will take memory, concentration, and thinking tests.
* Participants will have 3 MRI scans. An electroencephalography machine will record their brain activity. Electrodes will be placed on their scalp.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary objectives are to assess if there is an increase in the apparent diffusion coefficient (ADC) in the human brain during sleep when compared to the awake state and to determine if they vary across brain regions. Secondary outcomes are to assess inter subject variability in the differences in ADC between awake and sleep. We will also run exploratory analysis to determine if ADC changes with sleep are associated with subjective perception of rested sleep and to assess if there are differences in T1 in CSF between the scan taken prior to falling asleep and those taken shortly after waking up.

STUDY POPULATION:

Healthy adults. Males and females will be included.

DESIGN:

Observational study with a technical phase and two research phases.

* The technical phase (discontinued) will recruit controls in order to define best MR parameters and pulse sequence to be used for optimal ADC signal detection for which we request permission to recruit up to 20 healthy volunteers. Technical Developmental Phase: Each participant will have a set of MRI scans at the following two times of day: the 1st between 11:00 AM and 1:00 PM (noon) and the second between 6:00 PM and 8:00 PM (evening).
* Research Phase I (complete testing in 10 healthy controls to assess effects on wake/sleep states on whole brain ADC) and research Phase II (complete testing in a total of 30 subjects to assess if there are regional differences) and to address the main and secondary outcomes proposed above. Only if we show that ADC significantly changes during sleep compared to awake state will we proceed to phase II. For phases I and II, the participants will spend 3 night in the clinical center and will undergo two MRI scan sessions following two fo the night stays to quantify brain ADC; once while awake (following a night of sleep) and the other while asleep (following a night of sleep deprivation). Scans for both days will be performed in the morning (between 9-12 PM). Electrocardiogram (ECG) will be recorded during all MRI scanning procedures to monitor sleep. For the first of the three nights we will simultaneously record the electroencephalogram (EEG) and ECG on the participants while they sleep which will allow us to correlate the ECG to their EEG signal, which is the gold standard for measuring sleep.

OUTCOME PARAMETERS:

ADCs and ECG will be measured at each time point for each study participant (pertinent to research phase only).

ELIGIBILITY:
* INCLUSION CRITERIA:

All Participants

1. Between 18 and 60 years of age as determined by self-report.
2. Ability to provide written informed consent as determined by physical examination and verbal communication.

EXCLUSION CRITERIA:

All Participants

1. Subjects with self-report of insomnia as determined by self-report and/or medical history;
2. Subjects with any of the following: narcolepsy, obstructive sleep apnea (OSA) and/or abnormal sleeping patterns (including but not limited to those who use a C-PAP machine, sleeping during the day, using medication to fall asleep, sleeps less than 6 hours per night, night shift workers), subjects reporting snoring as determined by self-report using STOP-BANG questionnaire for undiagnosed OSA (3 or more yes answers will exclude) and/or medical history;
3. Subjects with a history of restless leg syndrome as determined by self-report and/or medical history;
4. Use, in the past two weeks, of psychoactive medications (four weeks for fluoxetine) or medications that may affect brain function (including but not limited to opioid analgesics, tricyclic antidepressants, selective serotonin reuptake inhibitors [SSRIs], or serotonin norepinephrine reuptake inhibitors [SNRIs], benzodiazepines and barbiturates) as determined by self-report and/or medical history;
5. Current or past DSM-IV or DSM 5 diagnosis of a psychiatric disorder as determined by history and clinical exam including substance use disorder (except for nicotine/caffeine), alcoholism and alcohol dependence. Past history of a mental disorder as defined by DSM IV or DSM 5 will be excluded only if it required hospitalization (any length), or chronic medication management (more than 4 weeks), and that could impact brain function at the time of the study.
6. Major medical problems that can impact brain function at the time of the scan (e.g., problems of the CNS including seizures and psychosis; cardiovascular disease including hypertension and arrhythmias; metabolic, autoimmune, endocrine disorders) as determined by self-report, medical history and/or clinical exam.
7. Head trauma with loss of consciousness for more than 30 minutes as determined by self-report and/or medical history;
8. Positive test for controlled substances (cocaine, methamphetamine, amphetamines, opioids, cannabinoids, benzodiazepines and barbiturates) on any day of study including upon check-in to NIH CC as determined by urine toxicology;
9. Pregnant: Females must have negative urine pregnancy test
10. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (including but not limited to pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces as determined by the self-report checklist.
11. Fear of enclosed spaces (claustrophobia) as determined by self-report and medical history.
12. Cannot lie comfortably flat on the back for up to 3 hours in the MRI scanner as determined by self-report.
13. Body weight greater than 250 kg. This is the upper limit that the bed of the MR scanner can accommodate (clinical exam).
14. Alcohol consumption on the day of the MRI as determined by breath alcohol test
15. Study investigators and staff, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
To assess if there is an increase in the apparent diffusion coefficient (ADC) in the human brain during sleep when compared to the awake state and to determine if they vary across brain regions. | end of study
  To assess if there are differences between brain regions.

SECONDARY OUTCOMES:
To assess inter subject variability in the differences in ADC between awake and sleep. | End of Study
  To determine if ADC differences are associated with subjective sense of rested sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Dardo G Tomasi, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Analysis is done in groups not on an individual basis.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-AA-0031.html